CLINICAL TRIAL: NCT05929560
Title: Diagnostic Evaluation and Guardian Assessment of Using Digital Impression in Neonates Versus the Conventional Techniques.
Brief Title: Digital Impression in Neonates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Hams Hamed Abdelrahman, Assistant lecturer of DPH and Clinical statistician, Alexandria University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Digital_impression_neonates_23
Record Dates: First submitted 2023-06-25; First posted 2023-07-03 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Unilateral Complete Cleft Lip and Palate

STUDY DESIGN:
Intervention Model Description: Paired design "Same patients receive conventional impression and digital"
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional impression (Active Comparator)
  Interventions: Other: Conventional impression
- Digital impression (Experimental)
  Interventions: Other: Digital impression

INTERVENTIONS:
Other: Conventional impression — Palatal impressions obtained using an irreversible hydrocolloid impression material
  Arms: Conventional impression
Other: Digital impression — after obtaining stone models from conventional impression material, stone models were scanned using the I700 (Medit) scanner and Patients were directly scanned intraorally using an intraoral 3D scanner Subsequently, the printed 3D model scan data of the seven patients were then used for standard triangulated language (STL)
  Arms: Digital impression

SUMMARY:
The goal of this [clinical trial] is to [explore the attitudes of guardians with different educational background regarding the technique of impression registration as well as the compliance to using feeding appliances ] in [neonates].

Researchers will compare [conventional impression technique to digital impression]

ELIGIBILITY:
Inclusion Criteria:

* patients with unilateral complete cleft lip and palate
* neonates

Exclusion Criteria:

* infants and children
* bilateral cleft lip and palatal
* incomplete cleft lip

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 7 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-06-15 (Actual)

PRIMARY OUTCOMES:
Deviation of linear measurments | up to 1 month
  The stone models obtained from conventional methods and 3D printed models obtained from the intraoral scanning were measured directly three times using an Vernier Fowler Calipers (WESTport Corporation, NY.),

SECONDARY OUTCOMES:
Assessment of gaurdian' perception and experience | up to 1 month
  The assessment of mothers' perception and experience regarding Pre-surgical infant orthopedics (PSIO) was executed using 16 validated preformed question.
  A questionnaire assess parents' satisfaction concerning PSIO

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria Faculty of Dentistry, Alexandria, Egypt